CLINICAL TRIAL: NCT06829784
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQC2731 Injections in Patients With Poorly Controlled Severe Asthma
Brief Title: TQC2731 Clinical Trial for the Treatment of Severe Asthma With Injection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2731-III-01
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC2731 injection (Experimental): TQC2731 injection, 4 weeks as a treatment cycle. Study drug administration from Day 0 up to Week 48.
  Interventions: Drug: TQC2731 injection
- Placebo (Placebo Comparator): Placebo,4 weeks as a treatment cycle.Study drug administration from Day 0 up to Week 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TQC2731 injection — TQC2731 injection can specifically bind to the Thymic Stromal Lymphopoietin (TSLP) protein, blocking TSLP-dependent downstream signaling expression in engineered cells and inhibiting the production of inflammatory cytokines.
  Arms: TQC2731 injection
Drug: Placebo — Placebo without drug substance.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel-group, placebo-controlled Phase III clinical trial designed to evaluate the efficacy and safety of TQC2731 injection (420 mg Q4W) in adult subjects with inadequately controlled severe asthma. A total of 660 subjects are expected to be enrolled, with subjects randomized in a 1:1 ratio to receive either TQC2731 (420 mg Q4W) or placebo (Q4W) via subcutaneous (SC) administration.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial to fully understand the purpose, process and possible adverse reactions of the trial;
* Age 18 ~ 75 years old, gender is not limited;
* Documented physician diagnosis of asthma at least 12 months prior to Visit 1;
* Subjects who received high-dose Inhaled Corticosteroids (ICS) in asthma control medications prescribed by their physicians at least 6 months prior to Visit 1;
* There must be a record of receiving a stable total daily dose of ICS at least 3 months prior to visit 1;
* There must be a record of the use of other asthma control medications at a stable dose at least 3 months prior to visit 1; For subjects taking maintenance oral hormones, the dose of oral hormones is up to 10mg prednisone per day or 20mg every other day (or equivalent) and must be stable for at least 30 days prior to visit 1 and during treatment.
* Documented at least 2 asthma exacerbations in the 12 months prior to Visit 1 and no major asthma exacerbation events in the 1 month prior to signing informed.

Exclusion Criteria:

* Have a clinically significant lung disease other than asthma；
* Pre-existing autoimmune disease;
* A history of known or suspected immunosuppression, including a history of invasive opportunistic infections;
* Any disease that has not been determined to be stable by the investigator；
* Cancer history: Patients with basal cell carcinoma, skin localized squamous cell carcinoma, or cervical carcinoma in situ are eligible to be enrolled in this study if they had completed curative therapy for at least 12 months prior to visit 1. Patients with other malignancies who had completed curative treatment for at least 5 years prior to visit 1 could be enrolled in the study.
* Current smoker or smoking history ≥10 pack-years (former smokers with smoking history <10 pack-years had quit smoking less than 6 months before interview 1);
* Other factors determined by the investigator that subjects were not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Annualized incidence of asthma exacerbations | From the first day of dosing to the completion of 52 weeks of treatment
  Annualized incidence of asthma exacerbations (AAER) during the 52-week treatment period.

SECONDARY OUTCOMES:
The change in forced expiratory volume in 1 second (FEV1) | Week 52 before dosing and before the use of bronchodilators (pre-Bronchodilator (pre-BD) administration)
  At Week 52, the change from baseline in forced expiratory volume in 1 second (FEV1) prior to dosing and before the use of a bronchodilator (pre-BD administration).
Change in total score of standardized asthma quality of life questionnaire | From baseline to week 52
  Change from baseline in standardized asthma quality of life questionnaire (AQLQ(S)+12) total score at week 52. Scores above 5 points indicate a relatively good quality of life, while scores below 3 points suggest a relatively poor quality of life.
Change in Asthma Control Questionnaire-6 (ACQ-6) score | From baseline to week 52
  Mean change from baseline in weekly mean asthma symptom diary score at week 52, , The higher the score, the more severe the asthma symptoms.
Mean change in weekly mean asthma symptom diary score | From baseline to week 52
  Mean change from baseline in weekly mean asthma symptom diary score at week 52
Change in European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire score | From baseline to week 52
  Change from baseline in European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire score at Week 52, a higher score indicates a better quality of life.
Change in mean rescue medication use, average peak expiratory flow rate (PEF) in the morning and night | From baseline to week 52
  Change from baseline in the average weekly dose of rescue medication and the average peak expiratory flow rate (PEF) per week in the morning and night, respectively
Changes in exhaled nitric oxide Fractional exhaled nitric oxide (FENO) (ppb), peripheral blood eosinophils, total serum Immunoglobulin E (IgE). | From baseline to week 52
  Change from baseline in exhaled nitric oxide FENO (ppb) at week 52.
Changes in peripheral blood eosinophils | From baseline to week 52
  Change from baseline in peripheral blood eosinophils at week 52.
Changes in total serum IgE | From baseline to week 52
  Change from baseline in total serum IgE at week 52.
Time to first asthma exacerbation | Baseline to week 64
  Time to first asthma exacerbation
Proportion of subjects with ≥1 asthma exacerbation | Baseline to week 64
  Proportion of subjects with ≥1 asthma exacerbation
Number of days of glucocorticoid use due to acute exacerbations | Baseline to week 64
  Number of days of glucocorticoid use due to acute exacerbations
Average amount of hormone used per acute exacerbation (prednisone equivalent) | Baseline to week 64
  Average amount of hormone used per acute exacerbation (prednisone equivalent)
Incidence of anti-drug antibodies (ADAs) in subjects | Baseline to week 64
  Immunogenicity: Incidence of anti-drug antibodies (ADAs) in subjects and their titers.
Incidence of neutralizing antibodies(NAB) in subjects | Baseline to week 64
  Immunogenicity: Incidence of neutralizing antibodies (NAB).

CONTACTS AND LOCATIONS:
Locations (74):
- China (74):
  - The People's Hospital of Bozhou, Bozhou, Anhui
  - Anhui Chest Hoispital, Hefei, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Third People's Hospital of Huizhou, Huizhou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Affiliated Hospital of Medical University, Guilin, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Cangzhou Hospital of Integrated TCM-WM·Hebei, Cangzhou, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Da Qing Long Nan Hospital, Daqing, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Qiqihar First People's Hospital, Qiqihar, Heilongjiang
  - The Second People's Hospital of Jiaozuo City, Jiaozuo, Henan
  - Luo Yang Dong Fang People's Hospital, Luoyang, Henan
  - Zhoukou Central hospital, Zhoukou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital (The First Affiliated Hospital of Hunan Normal University), Changsha, Hunan
  - Loudi central hospital, Loudi, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - The Second People Hospital's of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangsu University Affiliated Hospital, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin University Second Hospital, Changchun, Jilin
  - The First Hospital of Jlin University, Changchun, Jilin
  - Gansu Provincial Hospital, Gansu, Lanzhou
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Genertec Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - People's Liberation Army North Theater General Hospital, Shenyang, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical Universi, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - Affiliated Hospital of Jining Medical Hospital, Jining, Shandong
  - Weifang NO.2 People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Rui Jin Hospital Shanghai Jiaotong University School of Medical, Shanghai, Shanghai Municipality
  - Fudan University Affiliated Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Fudan University Affiliated Pudong Medical Center, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Wusong Central Hospital, Baoshan District, Shanghai, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Yangquan Coal Industry Group General Hospital, Yangquan, Shanxi
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin 4th Center Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xinjiang Uiger Municipal People'S Hospital, Ürümqi, Xinjiang
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The People's Hospital of Yuyao, Yuyao, Zhejaing
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Taizhou Central Hospital(Taizhou University Hospital), Taizhou, Zhejiang
  - Wenzhou Medical University Affiliated Second Hospital, Wenzhou, Zhejiang